CLINICAL TRIAL: NCT02299453
Title: Telephone IPT Intervention for HIV-Infected Rural Persons
Brief Title: Tele-IPT for HIV-Infected Rural Persons
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: Ohio University (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Timothy G. Heckman, Professor and Associate Dean for Research, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-10374
Record Dates: First submitted 2014-11-11; First posted 2014-11-24 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: HIV/AIDS; Depression
Keywords: Telemedicine; Interpersonal Psychotherapy (IPT)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants receive 9 sessions of telephone-administered PT and have access to standard community-based services. As part of the 9 sessions, participants discuss the extent to which interpersonal issues such as bereavements, role transitions, interpersonal disputes, and relationship difficulties may be related to their depression.
  Interventions: Behavioral: IPT
- Standard of Care (No Intervention): Participants receive no active intervention but do have access to standard community-based services, such as individual therapy, support groups, 12-step programs, and other social serves.

INTERVENTIONS:
Behavioral: IPT — Nine sessions of telephone-administered interpersonal psychotherapy (IPT)
  Arms: Experimental

SUMMARY:
This randomized clinical trial is testing if telephone-administered interpersonal psychotherapy (IPT) can reduce depression in rural persons living with HIV/AIDS.

DETAILED DESCRIPTION:
Compared to their urban counterparts, HIV-rural persons are more likely to be diagnosed with depression, less likely to seek assistance from mental health professionals, and appear to have shorter periods of survival. This application responds to PA-07-103 ("Research on Rural Mental Health and Drug Abuse Disorders") and the PA's stated need for research that will "Study whether individuals with various mental disorders can be treated effectively via telemedicine." A pilot RCT recently completed by our team showed that a 6-session telephone-delivered, interpersonal psychotherapy (IPT) intervention reduced depressive symptoms in 79 HIV- infected rural persons (Ransom, Heckman, et al., 2008, Psychiatric Services). This follow-up RCT will enroll 180 persons living with HIV/AIDS in rural counties in the United States who are diagnosed with depression via telephone interviews. Participants will complete self-administered surveys at pre-intervention, post- intervention, and 4- and 8-month follow-up that assess depressive symptoms (the primary outcome measure), interpersonal problems, social support, and ART adherence. Participants will also provide weekly data (for 41 weeks) via interactive voice response (IVR) systems that assess depressive symptoms (41 weeks) and therapeutic alliance (9 weeks). Ninety (n=90) participants will be randomly assigned to a 9-session, one-on- one, telephone-delivered, IPT intervention and 90 will be assigned to a usual care comparison group. Linear mixed models (LMM) will test if IPT participants report greater reductions in depressive symptoms compared to usual care controls. Analyses of reliable change will test if a greater proportion of IPT participants report clinically-significant reductions in depressive symptoms compared to usual care controls. Using weekly data collected via IVR systems, time series analyses will test if IPT participants report greater decreases in depressive symptoms over a 41-week follow-up period compared to usual care control. Mixed models analyses will assess the importance of therapeutic alliance in telephone-delivered IPT. Public Health Significance: This study will test if nine sessions of telephone-administered interpersonal psychotherapy can reduce depressive symptoms in HIV-infected rural persons, a group that is increasing in size and that experiences great difficulty accessing mental health support services.

ELIGIBILITY:
Inclusion Criteria:

* 18-plus years of age;
* a diagnosis of HIV infection or AIDS;
* residence in a county with a Department of Agriculture Rural-Urban Continuum Code of "6," "7," "8," or "9";
* a diagnosis of Major Depressive Disorder (MDD), Partial Remission of MDD, or Dysthymia based on the Mood Module of the "Primary Care Evaluation of Mental Disorders;
* the participant does not expect to leave his or her current place of rural residence within the next year; and
* provision of informed consent.

Exclusion Criteria:

* serious cognitive or neuropsychiatric impairment;
* being diagnosed with, or currently taking medications for, bipolar disorder;
* being diagnosed with, or currently taking medications for, psychotic disorder.

Min Age: 18 Years | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-12; Primary Completion 2014-11 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in depressive symptoms | Pre-Intervention, Post-Intervention(one week after completing the 9 week therapy), Four-Month Follow-Up, and Eight Month Follow-Up
  Self-administered surveys. Pre-intervention surveys are administered one week before therapy is initiated. Post-intervention surveys are administered one week after completing the 9 week therapy. Four-month follow-ups occur 4 months after the last therapy session and 8-month follow-ups are completed 8 months after the final therapy session. Control participants complete all four measures with their time-matched experimental participant.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heckman TG, Heckman BD, Anderson T, Lovejoy TI, Markowitz JC, Shen Y, Sutton M. Tele-Interpersonal Psychotherapy Acutely Reduces Depressive Symptoms in Depressed HIV-Infected Rural Persons: A Randomized Clinical Trial. Behav Med. 2017 Oct-Dec;43(4):285-295. doi: 10.1080/08964289.2016.1160025. Epub 2016 Apr 26. PMID 27115565
- [Derived] Heckman TG, Markowitz JC, Heckman BD, Woldu H, Anderson T, Lovejoy TI, Shen Y, Sutton M, Yarber W. A Randomized Clinical Trial Showing Persisting Reductions in Depressive Symptoms in HIV-Infected Rural Adults Following Brief Telephone-Administered Interpersonal Psychotherapy. Ann Behav Med. 2018 Mar 15;52(4):299-308. doi: 10.1093/abm/kax015. PMID 30084893